CLINICAL TRIAL: NCT05154422
Title: Differences in Lipolysis, Circulating Hormones, and Muscle Quality Between Recreational Female Endurance Athletes of Different Body Sizes
Brief Title: Effects of Regular Activity on Physiology Between Recreational Athletes of Different Body Fatness
Status: Completed | Type: Observational
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Principle Investigator, Florida State University
Other Study IDs: RALOW
Record Dates: First submitted 2021-01-26; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Obesity; Insulin Sensitivity
Keywords: Obesity; Muscle quality; Insulin Sensitivity; Lipolysis; Microdialysis; Endurance Training; Resistance Training; Exercise
MeSH Terms: conditions — Obesity; Insulin Resistance; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal body fat cohort: Determining the general amount of lipolysis, circulating insulin and growth hormone, and muscle quality of a group of recreational female endurance athletes with normal body fat determined by air displacement plethysmograph.
- Excess body fat cohort: Determining the general amount of lipolysis, circulating insulin and growth hormone, and muscle quality of a group of recreational female endurance athletes with excess body fat determined by air displacement plethysmograph.

SUMMARY:
The popularity of marathons and endurance events has increased over the last few decades and, interestingly, the demographics of participants have also changed. From 1980 to 2002 the average race time to complete the marathon lengthened from ~3.5 hours to ~4.5 hours. Likewise, many endurance races include "Clydesdale" and "Athena" divisions for heavier weight male and female runners, respectively. As such, there has been an increase of overweight and obese participants in these races. For example, one study consisting of 250 runners determined, according to BMI, that approximately 15% and 31% of the female and male participants, respectively, were classified as overweight, with 31% and 33% classified as obese. Therefore, many recreational endurance athletes are overweight despite their high level of activity. On one hand, these data are positive as regular exercise reduces cardiovascular disease and all-cause mortality in overweight and obese populations. Yet, it is well documented in sedentary obese individuals that excess adiposity can lead to disturbances in adipocyte lipolysis and altered substrate utilization at rest and during exercise, and can decrease muscle quality. However, it is unknown if overweight individuals that exercise regularly have disrupted fat metabolism, circulating hormones, or muscle quality. No study has directly determined if differences exist in fat metabolism, circulating hormones, and muscle quality between overweight recreational female athletes and their lean counterparts when training status is equivalent. Therefore, the purpose of this investigation is to determine if differences in pre and post-exercise fat metabolism, circulating insulin and growth hormone, and muscle quality exist between active overweight individuals compared to active lean individuals with similar training history and who have regularly trained for and participated in endurance events within the last few years.

DETAILED DESCRIPTION:
Fourteen active female endurance athletes (8 lower body fat, 6 higher body fat) will be recruited to participate in this study. The study will consist of two experimental days at the Institute of Sports Science and Medicine (ISSM) and the Sandels building at Florida State University. Participants will arrive at the laboratory in a fasted state for laboratory testing days. All participants will fill out a health history questionnaire, physical activity questionnaire, and sign the informed consent before any testing will be performed.

Testing Day 1:

For Day 1 of testing, participants will arrive in the morning at ISSM for informed consent, anthropometric testing, body composition, resting blood pressure, and fitness testing. All testing will be overseen by a certified strength and conditioning specialist.

Anthropometrics:

Anthropometric and body composition measurements will be assessed on the first day in the lab to ensure inclusion criteria are met. Height and weight will be measured with a wall-mounted stadiometer (SECA, Hamburg, Germany) and a digital scale (Detecto®, Webb City, MO, USA) respectively, and used to calculate body mass index (BMI: kg/m2). Fat-free mass, fat mass, and percent body fat will be assessed by Bod Pod (Cosmed, Chicago, IL) following the manufactures instructions.

Fitness Testing:

A submaximal YMCA cycle ergometer (Monarch, Kroons väg, Vansbro, Sverige) test will be used to assess the current fitness levels. In accordance with COVID-19 precautions, participants will be asked to complete the test on an ergometer outdoors of the ISSM laboratory and maintain PPE and social distancing as previously described. The test consists of three to four, three-minute stages. The first stage of the test starts with the participants pedaling against the resistance of 0.5 kg (150 kgm/min) at 50 rpm. Heart rate will be recorded at the end of each minute and if the second and third-minute measurements are within five beats of each other the researcher will adjust the resistance depending on the last heart rate recorded (<80 bpm = 2.5 kg, 80 - 90 bpm = 2.0 kg, 90 - 100 bpm = 1.5 kg, and >100 bpm = 1.0 kg). The participant will continue to pedal at 50 rpm through each of the stages and each stage following stage two will increase by 0.5 kg. The test concludes when two heart rate readings (between 110 and 150) have been collected in two different stages. The heart rate measurements and intensity for the two stages will be used to estimate the participant's VO2peak using the following equations: VO2max (ml/kg/min) = a (HRmax - HR2) + VO22, "a" is the slope of the line created by the HR and VO2 in the two stages of the test169. Before the test, participants will be fitted with a chest strap heart rate monitor and watch receiver (Polar, Lake Success, NY) which will continuously record the heart rate for the duration of the test. Participants will also be asked to rate their perceived exertion throughout the test. A Borg scale ranging from 6 to 20, 6 being equivalent to resting and 20 being equivalent to maximal effort, to determine how hard they felt they were working during the fitness test.

Compositional Muscle Quality Testing:

Following a standard 20-minute rest period, participants will be asked to sit on an examination table. Images of the rectus femoris will be taken midway between the inguinal crease and the proximal aspect of the patella using ultrasound. The intramuscular fat percentage of the rectus femoris will be assessed via analysis of the ultrasound echo intensity and related calculations. All parameters of the sonograph unit (depth, gain, etc.) will be kept constant between each participant. The average of the two measurements will be used to quantify echo intensity. Echo intensity of the measurements will be quantified via Adobe Photoshop histogram analysis (San Jose, CA) and will be used to estimate the intramuscular fat percentage using the following equations.

Females: y = [(0.062) • (40 • z + x)] + 7.901 Males: y = [(0.114) • (40 • z + x) + 1.126]

*x = raw echo intensity, y = intermuscular fat percent, z = subcutaneous adipose thickness

Functional Muscle Quality Testing:

Cross-sectional measurements of the rectus femoris (ultrasound measurements) with the isokinetic strength test will be used to calculate functional muscle quality (FMQ = N-m/mm2). Force production will be accessed via isokinetic dynamometry (Biodex Medical Systems Inc, Shirley, NY) using knee extension and flexion at 60º/s for strength testing. Participants will perform 2 sets of 3 reps, the peak power of the sets will be used as the measurement of maximal force production (N-m). A 2-minute rest will be given between sets. Isokinetic testing is not a usual mode of exercise as it requires equipment generally only found in a lab setting. Likewise, the specific test we will be conducting requires a very short period of time during physical exertion. The test does not increase minute ventilation, as it will take approximately 15 seconds per set for a total of 30 seconds of exercise. Therefore, this test will not increase the risk of COVID-19 spread. However, to reduce any possible risk of spreading COVID-19 participants will be required to wear a face-covering during this test, as well as social distancing protocols are being followed by the investigation team during the test.

7-Day Lifestyle Measurements At the end of the testing on this day, the participants will be given a packet with food and exercise logs, accelerometers (Actigraph WGT3X-BT, Pensacola, FL), and fatigue science bands (Vancouver, BC, Canada) to use over the following seven days. The information packet will also contain contact information to the research team in case a problem should arise with any of the equipment.

During the next 7 days, participants will keep track of their daily training routines by recording their distance, time to completion, and the rate of perceived exertion for the training session. They will wear an accelerometer (Actigraph WGT3X-BT, Pensacola, FL) to record their non-structured physical activity, and a fatigue science band (Vancouver, BC, Canada) to track sleep duration and quality.

Participants will also fill out food logs for all seven days for quantifying their normal diet. Information from the food logs will be analyzed (The Food Processor© Nutrition Analysis Software from ESHA Research, Salem, Oregon) for caloric and macronutrient (carbohydrate, protein and fat) content Training logs will be used by the participants to record their training sessions. The information recorded will be distance, duration, and session rate of perceived exertion. Accelerometers will be used to account for non-structured physical activity and quantify potential differences in sedentary time. Fatigue science bands will be used to record sleep quality, latency, and duration. All these parameters will be used to explore potential differences between the two groups and allow for potential covariate analyses.

Testing Day 2:

After the 7-day period of at-home data collection, participants will report back to the lab for the second day of testing (occurring no more the 10 days after day 1). Participants will arrive in the morning at the ISSM for microdialysis testing, metabolic measurements, exercise, and blood draws.

Lipolytic Response to Exercise:

Two microdialysis probes will be inserted percutaneously 5 - 10 cm lateral to the umbilicus for collection of interstitial glycerol for quantification of lipolysis. The microdialysis probes will be perfused with a solution of 0.9% sodium chloride and ~10 mM ethanol (for blood flow quantification) at 2.0 µL/min9,122. Interstitial glycerol concentration will be calculated via the following equation similar to other studies:

Gly in vivo = (Gly dialysate (1 - EtOH dialysate/perfusate) / (in vitro EtOH relative recovery / in vitro Gly relative recovery) After a 45-minute microdialysis probe equilibration period, resting dialysate will be collected for a total of 60 minutes (collection vials changed every 15 minutes). Next, participants will complete a 45-minute cycle ergometer (Velotron, Sram, Chicago, IL) ride (outside of the ISSM laboratory in open air) at 70% of their estimated VO2peak. Participants will be allowed to pedal at a conformable cadence as the ergometer will maintain watts despite RPMs. During the ride, participants will be given 125 ml of water every 15 minutes. One dialysate collection will occur immediately following the completion of the ride. Dialysate will then be collected for 120 minutes after physical activity (collection vials changed every 15 minutes). Participants will be allowed to sit up and read quietly in the lab for all post-physical activity data collection. Fat oxidation will be measured via indirect calorimetry for 30 minutes pre and immediately post-exercise, and again for the last 30 minutes of the 120-minute post-exercise. Dialysate will be stored at 4ºC for analysis of ethanol within 24 hrs. and subsequently stored at -80ºC until batch analysis of all dialysate glycerol samples (CMA600, Solna, Sweden).

Microdialysis Ethanol Outflow/Inflow Ratio

Ethanol (~10 mM) will be included with the perfusion medium to monitor adipose tissue blood flow in the area of the microdialysis probe9. Ethanol diffuses over the dialysis membrane and is not metabolized in adipose tissue to any significant extent. The Ethanol is transported away from the local area by the microcirculatory blood flow in the immediate vicinity of the probe membrane. An enzymatic fluorometric method is used to measurement the ethanol in the perfusate and dialysate. Blood flow will be expressed as a ratio of the ethanol concentration in the dialysate (outflow) and the ethanol concentration in the perfusate (inflow):

Ethanol outflow/inflow ratio = [ethanol dialysate]/[ethanol perfusate] The ethanol outflow/inflow ratio is inversely related to the local adipose tissue blood flow. Indirect calorimetry using a Parvo metabolic cart (TrueOne 2400; Parvomedics; Salt Lake City, UT) will be used to measure resting energy expenditure and determine whole-body fat oxidation at rest and post-exercise.

Metabolic Procedures and Exercise Stimulus Seventy-five minutes after insertion of the microdialysis probes, participants will be asked to lie in a supine position for 30 minutes to measure resting energy expenditure and respiratory exchange ratio, for quantification of whole-body fat oxidation at rest. Following resting metabolic measurements, participants will be escorted outside of the lab to the track. Participants will be instructed through a standardized dynamic warm-up lasting about five minutes (appendix A). The participants will then be instructed to ride on a monarch cycle ergometer maintaining 90 revolutions per minute for 45 minutes. The resistance will be set to elicit about 2 - 3 watts per kilogram of lean body mass, set to correspond with approximately 70% estimated VO2peak. In accordance with COVID-19 precautions, the warm-up and cycling will be performed while maintaining a safe and recommended social distance (at least 6 feet). Immediately after the cycling bout the participant will be escorted back into the lab and will be asked to lie down in a supine position for 30 minutes of continuous gas collection for measurement of post-exercise energy expenditure, respiratory exchange ratio, and fat oxidation. These measurements will be taken again in the same supine position for 30 minutes at the end of the 120-minute post-exercise period.

Circulating Hormone Changes to Exercise Venous blood samples, via an antecubital vein, will be collected to measure concentrations of insulin, human growth hormone, atrial natriuretic peptide, and glucose. A total of three blood draws will be collected, during the microdialysis testing day immediately before and after the exercise bout, as well as 120 minutes post-exercise. Plasma insulin and growth hormone will be compared between groups and used as a covariate for lipolytic action.

All blood will be collected in heparin-coated plasma vacutainers and will be centrifuged for 15 min at 3,500 rpm at 4 °C and aliquots plasma will be stored at -80°C for later batch analysis to limit day-to-day assay variability. Capillary blood glucose and HbA1c via a finger stick will be measured with a hand-held glucometer (OneTouch Ultra, LifeScan Europe, CH), and a DCA Vantage analyzer (Siemens, Tarrytown, NY), respectively. Plasma insulin (R&D systems, DINS00, Minneapolis, MN) and human growth hormone (R&D systems, DGH00, Minneapolis, MN) will be assessed via enzyme-linked immunosorbent assay according to the manufacturer's instructions. Blood will be drawn immediately following metabolic testing for resting measurements, immediately after the cycling bout, and at 120 minutes post-exercise.

ELIGIBILITY:
Inclusion Criteria:

* Female participants will be recruited for the study
* (BMI of <29.9 kg/m2).
* Ages of 18 and 45 years old
* Weight stable (± 2 kg) for the last three months
* Regularly endurance training on most days of the week for at least one hour for the last two years
* No exclusion will be made for race or socioeconomic status
* Participants will be eumenorrheic and premenopausal

Exclusion Criteria:

* Resting blood pressure above 160 mmHg systolic or 100 mmHg diastolic
* Type 1 or type 2 diabetes; 3)
* Other medical problems in which exercise is contraindicated
* chronic infections
* Diagnoses, signs, or symptoms of cardiovascular disease
* Respiratory disease
* Musculoskeletal disease
* Musculoskeletal injuries in the last six months that would prevent them from engaging in endurance training.
* Pregnant or lactating and must have a
* Irregular menstrual cycle
* Smoking
* Diagnosed eating disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fourteen active female endurance athletes (8 lower body fat, 6 higher body fat) will be recruited to participate in this study
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Lipolysis | Second experimental visit for a total of 6 hours
  Tested via microdialysis. Two probe inserted into the subcutaneous abdominal adipose tissue to collect glycerol molecules (byproduct of lipolysis).
Change in circulating insulin around an exercise bout | Second experimental visit - Pre-exercise, Immediately post-exercise, and 120-minutes post-exercise
  Insulin will be collected via blood draws. Blood will be drawn immediately following metabolic testing for resting measurements, immediately after the bout of physical activity, and every hour for 120 minutes' post activity.
Change in circulating growth hormone around an exercise bout | Second experimental visit - Pre-exercise, Immediately post-exercise, and 120-minutes post-exercise
  Growth hormone Insulin will be collected via blood draws. Blood will be drawn immediately following
Compositional Muscle Quality | First experimental visit - 15 minutes
  Intramuscular fat accumulation percentage will be measured and estimated using B-mode ultrasound echo intensity via histogram analysis and composition equations
Functional Muscle Quality | First experimental visit - 30 minutes
  Functional MQ is measured via force production (via Biodex) divided muscle size (via dual energy X-ray absorptiometry).

SECONDARY OUTCOMES:
Blood Sampling Analysis | Second experimental visit - Pre-exercise, immediately after the resting metabolic measurements
  Blood will be analyzed for glucose, and lipid profile. Blood will be drawn immediately following metabolic testing for resting measurements for these resting measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Science and Medicine, Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided